CLINICAL TRIAL: NCT06978387
Title: The Association Between Glycemic Metrics and Cardiovascular Markers in Patients With Type 1 Diabetes.
Status: Recruiting | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, VAIA LAMBADIARI, Professor of Internal Medicine-Endocrinology, Attikon Hospital
Other Study IDs: TYPE 1_CROSS-SECTIONAL
Record Dates: First submitted 2025-01-30; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Type 1 Diabetes Mellitus: patients aged >12 years old with T1DM who are on MiniMed 780G
  Interventions: Device: Minimed 780G

INTERVENTIONS:
Device: Minimed 780G — patients aged >12 years old with T1DM who are on MiniMed 780G

SUMMARY:
In this cross-sectioanl study, 90 patients aged >12 years old with T1DM who are on MiniMed 780G system will be included.The investigators aim to assesse the association of patients' adherence to Mediterranean diet (MD) with CGM and insulin metrics, as well as anthropometric measurements, BMI, lipid levels and blood pressure.Moreover, markers of endothelial, cardiovascular and liver function will be also assessed and associated with the use of Minimed 780G and the adherence to MD.

DETAILED DESCRIPTION:
This cross-sectional study will include 90 participants, children adolescents and young adults (12> years old) with T1D that are on MiniMed 780G system. Participants will be evaluated for adherence to Meditteranean Diet (MD) with PREDIMED questionnaire. HbA1c, CGM and Insulin Metrics, anthropometric measurements, blood pressure and lipid leves will be aso evalutaed. Markers of endothelial cardiovascular and liver function will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes >1 year prior to consent date. Diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not required.
2. HbA1c < 12.5%
3. Age >7years at the initiation of the system
4. Patients with Minimed 780G
5. History of 3 clinic visits in the last year

Exclusion Criteria:

Diabetic Ketoacidosis in the 6 months prior to screening visits

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children adolescents and young adults (12> years old) with T1D that are on MiniMed 780G system.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Time in Range | Baseline
  Assessment of time in range
Time below range | Baseline
  Assessment of time below range
Time above range | Baseline
  Assessment of time above range
Basal Insulin dose | Baseline
  Assessment of basal insulin doses
Correction Insulin dose | Baseline
  Assessment of correction insulin dose
Pulse wave velocity | Baseline
  Assessment of pulse wave velocity
Endothelial glycocalyx | Baseline
  Assessemnet of the thickness of endothelial glycocalyx
Global longitudinal strain | Baseline
  Assessment of global longitudinal strain.
E score | Baseline
  Assessement of E score and CAP score.
Assessment of CAP score | Baseline
  CAP score
MED diet | Baseline
  Assesment of Adherence to MED diet
Fat mass | Baseline
  Assessment of fat mass
Lean Mass | Baseline
  Assessment of lean mass

CONTACTS AND LOCATIONS:
Overall Officials: Vaia Lambadiari, Principal Investigator — Attikon General University Hospital
Locations (1):
- Attikon University General Hospital, Chaïdári, Greece